CLINICAL TRIAL: NCT03272958
Title: Clinical Characteristics of Pruritus and Evaluation of Quality of Life in Patients With Bullous Pemphigoid
Acronym: PRURIPB
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC17.0066 ( PRURIPB)
Record Dates: First submitted 2017-07-21; First posted 2017-09-06 (Actual); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Bullous Pemphigoid
Keywords: Pruritus; Bullous pemphigoid
MeSH Terms: conditions — Pemphigoid, Bullous; Pruritus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Whereas pruritus is a major symptom in bullous pemphigoid, its characteristics and its impact on quality of life have been little studied.

The objective of this study is to learn more about pruritus characteristics of patients with bullous pemphigoid, and in consequence to better understand the pathophysiology of pruritus, and then to better treat pruritus in this condition.

ELIGIBILITY:
Inclusion Criteria:

* adult
* pruriginous bullous pemphigoid lately diagnosed.
* Without PB treatment
* MMS (Mini Mental State Examination) ≥ 21
* In hospitalization or consultation

Exclusion Criteria:

* pregnant woman
* nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with a new diagnosis of bullous pemphigoid
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2018-10-03 (Actual); Study Completion 2018-10-03 (Actual)

PRIMARY OUTCOMES:
Clinical characteristics of pruritus in patients with bullous pemphigoid | Day1 ( when diagnosis of bullous pemphigoid is made)
  Answers and scores in questionnaire about clinical characteristics of pruritus Demographics characteristics of patients Characteristics of the bullous pemphigoid

SECONDARY OUTCOMES:
Impact of pruritus on quality of life in patients with bullous pemphigoid | Day 1 (when diagnosis of bullous pemphigoid is made )
  Score 5D itch scale
Impact of pruritus on quality of life in patients with bullous pemphigoid | Day1 (when diagnosis of bullous pemphigoid is made )
  score ItchyQol (Itchy Quality of Life)
Impact of pruritus on quality of life in patients with bullous pemphigoid | Day 1 (when diagnosis of bullous pemphigoid is made )
  score ABQOL

CONTACTS AND LOCATIONS:
Locations (16):
- France (16):
  - CH Argenteuil, Argenteuil
  - AP-HP, Hôpital Avicenne, Bobigny
  - CHU de Bordeaux, Bordeaux
  - CHRU de Brest, Brest
  - CHU Caen, Caen
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - AP-HP, Hôpital Henri Mondor, Créteil
  - CHU Le Havre, Le Havre
  - HP-HM, Marseille
  - CHU de Montpellier, Montpellier
  - CH de Niort, Niort
  - AP-HP, Hôpital Cochin, Paris
  - AP-HP, Hôpital Bichat, Paris
  - CHU de Reims, Reims
  - CHU de Rouen, Rouen
  - CHU de Saint-Etienne, Saint-Etienne